CLINICAL TRIAL: NCT05435508
Title: Efficacy in Reducing Anxiety, Stress, and Pain Levels Through Preanesthetic Assessment and Pain Neuroscience Education in Patients Undergoing Elective Total Abdominal Hysterectomy: A Randomized Clinical Trial
Brief Title: Efficacy of Pain Neuroscience Education and Pre-anesthetic Assessment in Reducing Levels of Anxiety, Stress and Pain in Patients Undergoing Elective Total Abdominal Hysterectomy (ENAH Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Neurociencia Del Dolor (Other)
Collaborators: Hospital Univeristario Benemerita Universidad Autonoma de Puebla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INeurocienciaDolor
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pain, Chronic; Pain, Postoperative; Anesthesia; Surgery; Anxiety; Stress
Keywords: Pain neuroscience education; Hysterectomy; Pre-anesthetic Assessment
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were blinded to group allocation. Care providers and the investigator delivering the intervention were not blinded due to the nature of the intervention. Data analysts remained blinded during statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Pain Neuroscience Education plus Pre-anesthetic Assessment (Experimental): Participants assigned to this arm received one face-to-face Pain Neuroscience Education (PNE) session (approximately 35 minutes) in addition to the standard pre-anesthetic assessment. PNE consisted of an educational intervention focused on the neurobiology and neurophysiology of pain and pain processing by the nervous system.
  Interventions: Other: Pain Neuroscience Education; Other: Usual care
- Pre-anesthetic Assessment (Usual Care) (Other): Participants assigned to this arm received standard pre-anesthetic assessment (usual care), which included evaluation of physical condition, medical and surgical history, and laboratory tests, in order to establish surgical risk and define the anesthetic plan according to the surgical procedure.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pain Neuroscience Education — One face-to-face Pain Neuroscience Education (PNE) session was delivered by a professional certified in PNE, with a duration of approximately 35 minutes. The session addressed the neurobiology and neurophysiology of pain, central sensitization, cortical representation of body regions, pain-related changes in body perception, and psychosocial dimensions of pain. Participants also received standard pre-anesthetic assessment, identical to the usual care group.
  Other Names: Therapeutic Neuroscience Education; Pain Neurophysiology Education
  Arms: Experimental: Pain Neuroscience Education plus Pre-anesthetic Assessment
Other: Usual care — Usual care consisted of standard pre-anesthetic assessment and routine perioperative management, including analgesic medication administered before, during, and after hysterectomy, according to institutional protocols and the clinical judgment of the attending physician.

SUMMARY:
Through this quantitative, multivariate factorial experimental parallel randomized clinical trial, the investigators analyzed the effectiveness of pre-anesthetic assessment and pain neuroscience education in reducing anxiety, stress, and pain levels in patients undergoing elective total abdominal hysterectomy.

DETAILED DESCRIPTION:
Hysterectomy is a common surgical procedure with a low risk of major complications. However, some women experience long-lasting complications, including chronic postsurgical pain, which can have a negative impact on their quality of life.

The population will be made up of women with elective total abdominal hysterectomy scheduled surgery at the University Hospital of Puebla BUAP, in the city of Puebla, Mexico.

Then the investigators will carry out an pre-anesthetic evaluation will be carried out and an pain neuroscience education session will be carried out.

Once patients are ready for surgery, the investigators will carry out an invasive monitoring will be performed in the post-anesthesia care unit. The blood pressure of the participants will be monitored non-invasively. They will also be monitored with electrocardiogram and pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

1. Anesthesia Physical Classification System: I, II or III according to the classification of the American Society of Anesthesiology.
2. Acceptance of informed consent
3. Basic literacy skills sufficient to understand and complete study questionnaires.

Exclusion Criteria:

1. Inability to understand study procedures or complete questionnaires.
2. Inflammatory rheumatic disease
3. Major neurological or psychiatric disease, Intellectual disability (mental retardation) or learning disorders at the premorbid level or severe language comprehension problems.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale-Pain (EVA) | Baseline (preoperative), 1 hour postoperative, and 8 hours postoperative
  Pain intensity at rest was assessed using a 10-cm visual analog scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
Change in Perceived Stress Scale - 14 items (PSS-14) | Baseline (preoperative), 1 hour postoperative, and 8 hours postoperative
  Perceived stress was assessed using the 14-item Perceived Stress Scale (PSS-14). Each item is rated on a 5-point Likert scale (0-4), yielding a total score ranging from 0 to 56, with higher scores indicating greater perceived stress.
Change in Beck Anxiety Inventory (BAI) | Baseline (preoperative), 1 hour postoperative, and 8 hours postoperative
  Anxiety symptoms were assessed using the Beck Anxiety Inventory (BAI), a 21-item self-reported questionnaire. Each item is scored from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate greater anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Johana Milena Mejía-Mejía, MD, Principal Investigator — Hospital Universitario de Puebla BUAP; Leidy Tatiana Ordoñez-Mora, MsC, Study Chair — Universidad Santiago de Cali, Cali, Colombia.; Michelle Dassaaejv Macias Amezcua, MD, Study Chair — Hospital Universitario de Puebla BUAP; Pedro Javier López-Perez, PhD, Study Chair — Universidad de la Costa, Barranquilla, Colombia; Marco Antonio Morales-Osorio, PhD, Study Director — Universidad Arturo Prat, Iquique, Chile.
Locations (1):
- Hospital Univeristario Benemerita Universidad Autonoma de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Result] Attias S, Keinan Boker L, Arnon Z, Ben-Arye E, Bar'am A, Sroka G, Matter I, Somri M, Schiff E. Effectiveness of integrating individualized and generic complementary medicine treatments with standard care versus standard care alone for reducing preoperative anxiety. J Clin Anesth. 2016 Mar;29:54-64. doi: 10.1016/j.jclinane.2015.10.017. Epub 2016 Feb 2. PMID 26897450
- [Result] Goudman L, Huysmans E, Ickmans K, Nijs J, Moens M, Putman K, Buyl R, Louw A, Logghe T, Coppieters I. A Modern Pain Neuroscience Approach in Patients Undergoing Surgery for Lumbar Radiculopathy: A Clinical Perspective. Phys Ther. 2019 Jul 1;99(7):933-945. doi: 10.1093/ptj/pzz053. PMID 30921465
- [Result] Brandsborg B, Nikolajsen L, Hansen CT, Kehlet H, Jensen TS. Risk factors for chronic pain after hysterectomy: a nationwide questionnaire and database study. Anesthesiology. 2007 May;106(5):1003-12. doi: 10.1097/01.anes.0000265161.39932.e8. PMID 17457133
- [Result] Gursoy A, Candas B, Guner S, Yilmaz S. Preoperative Stress: An Operating Room Nurse Intervention Assessment. J Perianesth Nurs. 2016 Dec;31(6):495-503. doi: 10.1016/j.jopan.2015.08.011. Epub 2016 May 6. PMID 27931701
- [Result] Ordonez-Mora LT, Morales-Osorio MA, Rosero ID. Effectiveness of Interventions Based on Pain Neuroscience Education on Pain and Psychosocial Variables for Osteoarthritis: A Systematic Review. Int J Environ Res Public Health. 2022 Feb 23;19(5):2559. doi: 10.3390/ijerph19052559. PMID 35270250
- [Derived] Morales-Osorio MA, Mejia-Mejia J, Calva Maldonado M, Pablo Yanez JC, Ordonez-Mora LT. Efficacy of preanesthetic assessment combined with pain neuroscience education in reducing anxiety, stress, and pain in elective hysterectomy: A randomized controlled trial protocol. Medwave. 2025 Oct 13;25(9):e3092. doi: 10.5867/medwave.2025.09.3092. PMID 41082712